CLINICAL TRIAL: NCT07341269
Title: Prospective Evaluation of the Effect of Different Intervals Between Extracorporeal Shock Wave Lithotripsy (ESWL) Sessions on Potential Renal Injury Using Urinary NGAL and KIM-1 Biomarkers
Brief Title: Urinary NGAL and KIM-1 After ESWL
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MAR.UAD.0027
Record Dates: First submitted 2025-12-20; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Urinary Stone; Renal Injury
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary NGAL and KIM-1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing extracorporeal shock wave lithotripsy (SWL)
  Interventions: Other: No Interventions; Other: No intervention

INTERVENTIONS:
Other: No Interventions — No study-specific intervention; patients receive standard-of-care SWL.
Other: No intervention — No study-specific intervention; patients receive standard-of-care SWL.

SUMMARY:
The goal of this prospective observational study is to evaluate the effect of different time intervals between extracorporeal shock wave lithotripsy (ESWL) sessions on renal injury using urinary biomarkers in patients with urinary system stone disease.

The main questions it aims to answer are:

Does the interval between consecutive ESWL sessions affect the degree of renal injury?

Are urinary NGAL and KIM-1 levels reliable biomarkers for detecting ESWL-related renal damage?

What is the optimal time interval between ESWL sessions to minimize renal injury?

If there is a comparison group, researchers will compare patients undergoing ESWL with different inter-session time intervals to determine whether shorter or longer intervals are associated with higher levels of renal injury biomarkers.

Participants will:

Undergo ESWL treatment for urinary system stones

Be assigned to one of two groups based on the time interval between ESWL sessions

Provide urine samples before ESWL and after three ESWL sessions

Have urinary NGAL and KIM-1 levels measured to assess renal injury

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Patients with an indication for extracorporeal shock wave lithotripsy (SWL) for urinary system stone disease

Exclusion Criteria:

* Positive nitrite on urinalysis prior to SWL
* Positive urine culture prior to SWL, defined as >10⁵ CFU/mL bacterial growth
* Suspected struvite stone, based on previous or partial stone analysis
* Presence of a nephrostomy tube
* Presence of urinary diversion
* History of bleeding disorders
* Pregnancy
* Use of anticoagulant therapy
* History of cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older with urinary system stone disease who are undergoing extracorporeal shock wave lithotripsy (SWL) as part of routine clinical care. Participants are prospectively observed to evaluate changes in urinary NGAL and KIM-1 levels as biomarkers of renal injury associated with SWL. Patients with active urinary tract infection, suspected struvite stones, urinary diversion, nephrostomy tube, bleeding disorders, pregnancy, anticoagulant use, or cardiac arrhythmia are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Change in urinary NGAL level | Within 2 weeks after completion of the third SWL session
  Difference in urinary NGAL levels measured before SWL and after completion of three SWL sessions
Change in urinary KIM-1 levels | Within 2 weeks after completion of the third SWL session
  Difference in urinary KIM-1 levels measured before SWL and after completion of three SWL sessions

SECONDARY OUTCOMES:
Between-group difference in change of urinary NGAL and KIM-1 levels according to SWL session intervals | Within 2 weeks after completion of the third SWL session

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine Urology Department, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No